CLINICAL TRIAL: NCT06584357
Title: Development of a Database to Investigate Digital and Blood-Based Biomarkers and Their Relationship to Tau and Amyloid PET Imaging in Older Participants Who Are Cognitively Normal (CN), Have Mild Cognitive Impairment (MCI), or Have Mild-to-Moderate AD Dementia
Acronym: Bio-Hermes-002
Status: Recruiting | Type: Observational
Sponsor: GAP Innovations, PBC (Industry)
Responsible Party: Sponsor
Other Study IDs: Bio-Hermes-002
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Alzheimer's Disease, Early Onset; Memory Loss; Memory Disorders; Memory Impairment
Keywords: Alzheimer's Disease; Alzheimer's Disease, Early Onset; Mild Cognitive Impairment; Older Volunteers; Healthy Volunteers; Memory Loss; Memory Disorders; Memory Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders | interventions — MK-6240

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * LucentAD
  * APOE
  * Aβ 42/40
  * p-tau 181/217/231
  * Total tau
  * NfL
  * Genome sequencing
  * Proteomics
  * Photonics
  * Other measures of neuroinflammation: GFAP, YKL-40, MCP-1, Factor B, Factor H, sCRI, Eotaxin, TNFα, CD8+T effector memory cells, DNases and RNases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitively Normal: No reported memory loss or concerns as reported by participant and study partner.
  Interventions: Other: Biomarker Data Collection; Radiation: MK6240
- Mild Cognitive Impairment: A diagnosis of Mild Cognitive Impairment (MCI) based on the National Institute of Aging (NIA) criteria and verified through medical records.
  Interventions: Other: Biomarker Data Collection; Radiation: MK6240
- Mild-to-Moderate AD Dementia: A diagnosis of Mild-to-Moderate AD Dementia based on the National Institute of Aging (NIA) criteria and verified through medical records.
  Interventions: Other: Biomarker Data Collection; Radiation: MK6240

INTERVENTIONS:
Other: Biomarker Data Collection — During this study, a sample of your blood will be collected and you will have a PET scan taken of your brain. Blood sample results will be compared to PET scan pictures to understand how well the markers in the blood predict whether there is amyloid in the brain. Blood samples will also be collected that contain your genes. These genetic samples will also be compared to PET scans to help researchers understand how different people react to medicines and to understand the genetic causes of AD. Some of the samples will be stored for future analysis.
Radiation: MK6240 — Each participant will be assessed using either one of two radioactive tau PET tracers: Flortaucipir or MK6240. Flortaucipir is FDA approved while MK6240 is not and is being used in this study as an investigational radioactive drug.

SUMMARY:
Bio-Hermes-002 is a 120-day cross-sectional study that will result in a blood, CSF, retinal, digital, MRI, and PET brain imaging biomarker database that can be used to determine the primary objective. Digital biomarkers and blood-based biomarkers will be tested to determine whether a meaningful relationship exists between biomarkers alone or in combination with tau or amyloid brain pathology identified through PET images.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening Inclusion Criteria

Participants must meet ALL of the following criteria to progress to Visit 1 (Screening):

1. Participant is between 60 to 90 years of age (inclusive) at the time of consent; and
2. Participant has a study partner who has sufficient and frequent contact with the participant (defined as at least 8 hours of contact a week) and is able to provide accurate information regarding the participant's cognitive and functional abilities.

Core Study Inclusion Criteria

Participants must meet ALL of the following criteria, in addition to the Pre-screening Inclusion Criteria, for entry into the study:

1. Participants must provide written consent in the IRB-approved or Ethics Committee (EC) approved informed consent form or have a legally authorized representative (LAR) provide written consent on the participant's behalf in accordance with local and national guidance and regulation;
2. Participants must be willing to undergo an MRI brain scan within 90 days and an amyloid and tau PET scan within 120 days of signing informed consent;
3. Participants must be willing to comply with all study procedures as outlined in the informed consent, including blood sampling, genetic testing, and storage of biospecimens for future research;
4. Fluency in the language of the tests used at the study site;
5. Participants must be willing to be contacted for possible participation in clinical research trials once their participation in this study ends; and
6. Participants must have a Mini-Mental State Exam (MMSE) score of 16 to 30 inclusive at screening.

Exclusion Criteria:

Pre-screening Exclusion Criteria

Participants who meet ANY of the following criteria will not be eligible to progress to Visit 1 (Screening):

1. Participant is unable to undergo amyloid and tau PET scans due to self-reported pregnancy, sensitivity to ligands being used, poor venous access, contraindication to PET, or planned or recent exposure to ionizing radiation that in combination with the planned administration of amyloid radioligand would result in a cumulative exposure that exceeds recommended local guidelines;
2. Participants who have reported or have a known negative amyloid PET scan in the past 6 months;
3. Participants with any known contraindication to brain MRI scan;
4. Participants with history of stroke or seizures within 1 year of the Pre-Screening Visit;
5. Participants with history of cancer within the past 5 years with the exception of non-melanoma skin cancer or prostate cancer in situ;
6. Participants with known or suspected alcohol or drug abuse or dependence within 1 year of the Pre- Screening Visit;
7. Participants who report any current unstable psychiatric symptoms that could interfere with study procedures or impact study data (e.g., uncontrolled depression);
8. Participants who have received any potential disease modifying AD treatment within 6 months prior to the Pre-screening Visit; and
9. Participants with known history or self-report to be Human Immunodeficiency Virus (HIV) Positive unless controlled by antiviral medication.

Core Study Exclusion Criteria

Participants who meet ANY of the following criteria, in addition to the Pre-screening Exclusion Criteria, will not be eligible to enroll into the study:

1. Participants who, in the opinion of the Site Principal Investigator, have serious or unstable medical conditions that would prohibit their completion of all study procedures and data collection;
2. Participants who have serious or unstable medical conditions that would likely preclude their participation in an interventional research trial;
3. Participants with self-reported, untreated conditions such as vitamin B12 or folate deficiency or bladder infections that in the opinion of the Site Principal Investigator could contribute to cognitive impairment;
4. Participants who have completed cognitive testing within 1 month of Visit 1 (Screening) where the Site Principal Investigator believes the participant's exposure may cause practice effect;
5. Participants who have any neurological disorder affecting the central nervous system, other than AD, that may be contributing to cognitive impairment (e.g., Parkinson's disease, other dementias, multiple concussions or seizures) as deemed significant by the Site Principal Investigator;
6. Participants with a Geriatric Depression Scale (GDS) score greater than or equal to 8 at Visit 1 (Screening) and is deemed to be clinically significantly depressed by the Site Principal Investigator;
7. Participants with a Rey Auditory Verbal Learning Test (RAVLT) t-score of ≥ 1.2 standard deviation above the mean. For non-African Americans, calculate age-sex-education adjusted t-scores. For African American participants, use the MOANS to calculate the age-education adjusted t-scores;
8. Participants weighing less than 110 pounds;
9. Participants who are direct employees or family members of direct employees of the participating investigators' sites;
10. Participants who are direct employees of the Sponsor;
11. Participants who, in the opinion of the investigator, are unable to complete cognitive testing due to inadequate visual or auditory acuity; and
12. For participants completing the RetiSpec retinal scan: Those with a known history of contraindication or allergy to Tropicamide 1% (pupil dilation drop).

Longitudinal Sub-Study Eligibility

Inclusion Criteria:

Participants must meet ALL of the following criteria for entry into the sub-study:

1. Participants who completed the Bio-Hermes-002 Core Study;
2. Are willing to complete phone call visits with site staff every three months and return to the clinic for an annual evaluation; and
3. Are willing to complete annual PET scans for both amyloid and tau scans.

Exclusion Criteria:

Participants who meet ANY of the following criteria will not be eligible for entry into the sub-study:

1. Those who are enrolled or intend to enroll into a clinical trial for Alzheimer's disease with a potential disease-modifying intervention;
2. Participants who have serious or unstable medical conditions that would likely preclude their participation in an interventional research trial;
3. Those who intend to use medications outside clinical research studies approved by regulatory authorities to modify Alzheimer's disease pathology.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 1,200 participants will complete all the activities of the protocol over an 18-month competitive enrollment period. Each site will be expected to enroll approximately 40 participants. Approximately 25% of the total participants enrolled will be from underrepresented populations. Enrolled participants will be characterized as fitting into one of three cohorts with approximately 1/3 enrollment in each cohort. While we have outlined cohort criteria below, ultimately it is up to the site principal investigator to determine cohort placement.
  Cohort status will not be shared with participants.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and PET | Through study completion, an average of 3 years
  Measure blood biomarkers (Aβ 42/40, p-tau 181, p-tau 217, p-tau 231, total tau, and NFL) to see if it will predict the extent of tau and amyloid brain pathology as measured by PET brain imaging in participants shown to be cognitively normal (CN), have mild cognitive impairment (MCI), or have mild-to-moderate AD dementia.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (22):
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - K2 - Winter Garden, Clermont, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of SW Florida, Fort Myers, Florida
  - K2 Medical Research, Maitland, Florida
  - Clincloud, Melbourne, Florida
  - Visionary Investigators Network, Miami, Florida
  - Charter Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Inc., Sarasota, Florida
  - Axiom Brain Health, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Flourish Research - Chicago, Chicago, Illinois
  - Quest Research Institute, Farmington Hills, Michigan
  - Clinical Neurology Specialists, Las Vegas, Nevada
  - ADRC of Albany, Albany, New York
  - Neuro-Behavioral Clinical Research Inc., North Canton, Ohio
  - Flourish Research - Philadelphia, Philadelphia, Pennsylvania
  - K2 Medical Research, East Providence, Rhode Island
  - Gadolin Research LLC, Beaumont, Texas
  - Re:Cognition Health, Houston, Texas
- Toronto Memory Program, Toronto, Ontario, Canada
- United Kingdom (2):
  - NeuroClin Glasgow, Motherwell, North Lanarkshire
  - Re:Cognition Health, London

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared but the plan has not been finalized.